CLINICAL TRIAL: NCT05368298
Title: Sample Collection for The Integration and Analysis of Data Using Artificial Intelligence to Improve Patient Outcomes With Thoracic Diseases
Brief Title: SCOOT: Sample Collection for DART
Acronym: SCOOT
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Innovate UK (Other Government); Optellum (Unknown); National Institute for Health Research, United Kingdom (Other Government); Cancer Research UK (Other); GE Healthcare (Industry); Prenostics (Unknown); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: OCTO-106
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: screening; lung health check; artificial intelligence; algorithm; diagnosis; detection
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — 30ml blood sample will be collected and processed, resulting in plasma and serum samples for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will use a blood sample collected from participants to:

* Develop new ways of finding and diagnosing lung health problems, such as lung cancer.
* Develop tools which make it easier to screen people with possible lung health problems, diagnose problems earlier and with fewer tests, and start the best treatment faster.
* Help improve the early diagnosis of lung cancer, as finding lung cancer early means that it can be treated more easily and successfully.

DETAILED DESCRIPTION:
The results from this study will be linked with the data from the DART study (also collecting data through the Lung Health Check programme) to develop new ways of using computer technology (artificial intelligence) to improve lung health care. The studies use computer programs (called 'algorithms') which can be trained to analyse medical samples. Once developed, these algorithms can be used to support doctors by increasing their speed and accuracy of diagnosing issues.

ELIGIBILITY:
Patient suitability will be assessed against the below criteria by the clinical teams managing the patients.

Inclusion Criteria:

1. Patients with a pulmonary nodule or nodule(s) detected on a CT scan performed as part of Lung Cancer Screening from the Lung Health Check centres, that require further investigation with a PET-CT scan, and / or biopsy, and / or resection
2. Willing and able to give informed consent

Exclusion Criteria:

* None -

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been offered follow up appointments after their Lung Health Check. Patients may be invited to attend a Lung Health Check if they have ever smoked and are aged 55 - 75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop an algorithm that gives a greater than chance improved ability to diagnose lung cancer using the blood biomarkers with or without the AI CT algorithm compared to not using them | by February 2025

SECONDARY OUTCOMES:
To develop an algorithm that gives a greater than chance improved ability to diagnose lung cancer using the blood biomarkers with or without the AI CT and blood markers algorithm compared to not using them | by February 2025

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Lung Health Check: Oxford - Churchill Hospital, OUH, Oxford, Oxfordshire
  - Lung Health Check Centre: Royal Sussex, Brighton
  - Lung Health Check Centre: North Bristol, Bristol
  - Lung Health Check Centre: Gateshead, Gateshead
  - Lung Health Check Centre: Corby & Kettering, Kettering
  - Lung Health Check Centre: Cheshire & Merseyside, Liverpool
  - Lung Health Check Centre: RM Partners, London
  - Lung Health Check Centre: Newcastle & Gateshead, Newcastle
  - Lung Health Check Centre: Plymouth, Plymouth
  - Lung Health Check Centre: Stoke, Stoke
  - Lung Health Check Centre: South Tyneside and Sunderland, Sunderland

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plans for the current study are unknown and will be made available at a later date.

REFERENCES:
- See also: OCTO webpage containing information about the SCOOT trial — https://www.oncology.ox.ac.uk/clinical-trials/oncology-clinical-trials-office-octo/prospective-trials/scoot
- See also: Cancer Research UK webpage containing information about the Lung Health Check programme — https://www.cancerresearchuk.org/about-cancer/lung-cancer/getting-diagnosed/lung-health-checks